CLINICAL TRIAL: NCT05873868
Title: MyocardON-TTR - Myocardial Effects in Patients With Hereditary Transthyretin-mediated Amyloidosis With Polyneuropathy Treated With Patisiran or Vutrisiran
Brief Title: Myocardial Effects in Patients With ATTRv With Polyneuropathy Treated With Patisiran or Vutrisiran
Acronym: MyocardON-TTR
Status: Active, not recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC22_9817_MyocardON-TTR
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloidosis; Amyloidosis, Hereditary
Keywords: Patisiran; Vutrisiran
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients hATTR with neurological and cardiac damages treated with Patisiran or Vutrisiran
  Interventions: Other: Six minutes walk test; Other: Kansas City questionnaire; Other: COMPASS31 self questionnaire

INTERVENTIONS:
Other: Six minutes walk test — Six minutes walk test just before first intake of treatment and after 1 and 2 years
Other: Kansas City questionnaire — Kansas City questionnaire just before first intake of treatment and after 1 and 2 years
Other: COMPASS31 self questionnaire — Compass31 self questionnaire assessing dysautonomia just before first intake of treatment and after 1 and 2 years

SUMMARY:
ATTRv amyloidosis is a systemic disease with two clinical forms, neurological and cardiological, which are sometimes combined (so-called mixed forms).

Patisiran and vutrisiran have shown protective effects on the progression of neurological damage.

The effects of Patisiran or vutrisiran on the heart remain incompletely understood. The aim of this study is to better understand the morphological and functional cardiac consequences in ATTRv patients with stage 1 or 2 polyneuropathy with a mixed form treated with Patisiran or vutrisiran

DETAILED DESCRIPTION:
ATTRv amyloidosis is a systemic disease with two clinical forms, neurological and cardiological, which are sometimes combined (so-called mixed forms).

Patisiran and vutrisiran have shown protective effects on the progression of neurological damage.

The effects of Patisiran or vutrisiran on the heart remain incompletely understood.

During their therapeutic management, including the prescription of Patisiran or vutrisiran, the routine examinations carried out at the inclusion, one and two year later will allow us to observe the consequences on myocardial activity during the routine consultation after 1 and 2 years of treatment.

Examinations are : clinical and biological exams, EKC, echocardiography, cardiac MRI and scintigraphy.

Data at the start of treatment and at 1 and 2 years will be collected, especially cardiac function assesment In addition, during these two consultations, a life quality questionnaire, a dysautonomia questionnaire and a functional walking test will be carried out specifically for the study.

The aim of this study is to better understand the morphological and functional cardiac consequences in ATTRv patients with stage 1 or 2 polyneuropathy with a mixed form treated with Patisiran or vutrisiran.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with hereditary transthyretin amyloidosis (ATTRv) with stage 1 or 2 polyneuropathy
* Patient not previously treated for ATTRv
* Patients for whom treatment with patisiran or vutrisiran has been initiated by a hospital neurologist in accordance with recommendations for a minimum of 24 months.
* Patients with NYHA stage 1 and 2 cardiac disease.
* Beneficiary of a social security scheme
* Person who does not object to his/her participation in the research

Exclusion Criteria:

* Patients treated with Tafamidis simultaneously with patisiran or vutrisiran
* Adults under legal protection (legal guardianship, curatorship, guardianship), persons deprived of liberty.
* Contraindications to the explorations provided for in the protocol: claustrophobia, metallic implant contraindicating MRI, woman of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hereditary transthyretin amyloidosis (ATTRv) with stage 1 or 2 polyneuropathy treated with Patisiran or Vutrisiran
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Difference in longitudinal relaxation time (T1) per mapping between M0 and M24 | 24 months
  Longitudinal relaxation time (T1) is the process by which the net magnetization (M) grows/returns to its initial maximum value (Mo) parallel to Bo in a MRI.
  Myocardial T1 depends on the pulse sequence, cardiac cycle as well as other factors and increases at higher magnetic field strength. T1-mapping can detect a variety of myocardial pathologies, where it shows increased values. Because of variations between scanners the primary use of a local reference range is recommended and if a local reference range is not available quantitative results should not be clinically reported. An intermediate analysis will be done at 12 months

SECONDARY OUTCOMES:
Difference in Kansas City Cardiomyopathy Questionnaire score between M0 and M24 | 24 months
  Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life. Five scores are generated, all scores are scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest. An intermediate analysis will be done at 12 months
Difference in Compass31 questionnaire score between M0 and M24 | 24 months
  The COMPASS-31 (Composite Autonomic Symptom Score-31) scale measures neurodegenerative system symptoms through 31 patient-reported questions. Assessment is through six weighted domains: orthostatic intolerance [10 points]; vasomotor [6 points]; secretomotor [7 points]; gastrointestinal [28 points]; bladder [9 points] and pupillomotor [15 points]. A higher score indicates worse autonomic dysfunction. An intermediate analysis will be done at 12 months
Difference in distance obtained in the 6-minute walking test between M0 and M24 | 24 months
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meter covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An intermediate analysis will be done at 12 months
Difference in Perugini Grading Score between M0 and M24 | 24 months
  The Perugini grading scale is a semi-quantitative method of scoring cardiac uptake following injection of 99mTc-DPD, 99mTc-Pyrophosphate or 99mTc-HMDP scintigraphy in the investigation of cardiac amyloidosis (particularly ATTR amyloidosis). The grading scale visually compares tracer uptake in the myocardium and ribs.
  grade 0 is no cardiac and normal rib uptake; grade 1 is cardiac less than rib uptake; grade 2 is cardiac equal to rib uptake; and grade 3 is cardiac greater than rib uptake with mild/absent rib uptake. An intermediate analysis will be done at 12 months
Difference in the value of the global longitudinal strain between M0 and M24 | 24 months
  global longitudinal strain is a simple parameter in echocardiography to analyse atrial function abnormalities expressed in percentage that expresses longitudinal shortening as a percentage (change in length as a proportion to baseline length) for left ventricular (LV) systolic dysfunction. An intermediate analysis will be done at 12 months
Difference in the value of the global left atrial longitudinal strain between M0 and M24 | 24 months
  Global left atrial longitudinal strain is a parameter of echocardiography to analyse atrial function abnormalities expressed in percentage. An intermediate analysis will be done at 12 months
Difference in the value of the global strain of the right ventricular free wall between M0 and M124 | 24 months
  Global strain of the right ventricular free wall of echocardiography to analyse right ventricule function expressed in percentage. An intermediate analysis will be done at 12 months
Evolution of myocardial work between M0 and M24 | 24 months
  Myocardial work is composed of 4 parameters to assess myocardial function using echocardiography. An intermediate analysis will be done at 12 months
  Global Constructive Work (expressed in mmHg%) : Positive work performed in systole (shortening) + Negative work performed in isovolumetric relaxation (lengthening). Normal range : 1582-2881
  Global Wasted Work (expressed in mmHg%) : Negative work performed in systole (lengthening) + Positive work performed in isovolumetric relaxation (shortening). Normal range : 226 ± 28
  Global Work Efficiency (expressed in %) Percentage (0-100%) of constructive work over total work => Constructive work/(constructive work + wasted work). Normal range : 91 ± 0.8
  Global Work Index (expressed in mmHg%) : Amount of myocardial work performed by the left ventricle during systole => area of PSL from mitral valve closure to mitral valve opening. Normal range : 1292-2505

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - CHU Bordeaux Haut-Levêque, Bordeaux
  - APHP Henri Mondor, Créteil
  - CHU Grenoble Alpes, Grenoble
  - CHU Nancy Institut Louis Mathieu, Nancy
  - CHU Rangueil Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided